CLINICAL TRIAL: NCT05951257
Title: Feasibility and Efficacy of Hypnosis and Music on Pain, Anxiety and Well-being in End-of-life Palliative Care at Home
Brief Title: Medical Hypnosis and Music for Palliative Care
Acronym: MuzhypforPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Principal Investigator, Josiane Bissonnette, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MP-23-2022-896
Record Dates: First submitted 2023-07-03; First posted 2023-07-19 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Palliative Care; Pain Management; Anxiety; Well-being
Keywords: Hypnosis; Music
MeSH Terms: conditions — Agnosia; Anxiety Disorders | interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: Experimental group: 2 intervention sessions ; Control group (waiting list): 2 control sessions followed by 2 intervention sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized multimodal intervention involving hypnosis and/or music (Experimental): This arm will receive a personalized multimodal intervention involving (a) hypnosis, (b) music or (c) hypnosis and music.
  Note that the objective of the research is not to compare the effect of the different intervention modalities between them, but to consider these three modalities as a multimodal intervention taking into consideration patients' preferences, that we compare to the control.
  Interventions: Behavioral: Personalized multimodal intervention involving hypnosis and/or music
- Control/Waiting list (No Intervention): The participants of the control group will carry out its their daily activities and will be assessed using the same measures, at the beginning of each session and after a delay comparable to the duration of the intervention administered in the experimental group.

INTERVENTIONS:
Behavioral: Personalized multimodal intervention involving hypnosis and/or music — The three intervention modalities (music and/or hypnosis) will begin by a moment of relaxation in which we will ask the participants to focus their attention on their breathing, on relaxation and on the process of absorption into oneself. The hypnosis modality consists in visiting in imagination a pleasant place that the participant will choose and to live some metaphorical stories. The "musical" modality consists of listening to one or two pieces of music chosen by each participant and which brings him/her well-being, according to them. These two types of work will be preceded by a moment of relaxation in which we will ask the participants to focus their attention on their breathing, on relaxation and on the process of absorption into oneself.
  Other Names: MuzHyp program; Hypnosis and music intervention program
  Arms: Personalized multimodal intervention involving hypnosis and/or music

SUMMARY:
The goal of this randomized controlled trial is to evaluate the efficacy of a personalized multimodal intervention program (MuzHyp) including hypnosis, music or their combination to improve palliative care at home.

The main objective is to evaluate if the intervention program will significantly reduce participants' composite score of pain, anxiety, and unwellness as evaluated by the Edmonton symptom assessment scale (ESAS) immediately after the intervention, and whether this improvement will be significantly greater than that of control sessions.

DETAILED DESCRIPTION:
Context :

Quality of life at home in end-of-life palliative care is an ideal that is often difficult to achieve. Side effects of medications and limited access to resources and services can affect the control of pain, anxiety and well-being. Research shows that musical interventions and the use of medical hypnosis can help reduce pain and anxiety, and thus improve patients' psychological well-being in many clinical settings. In view of this, we have developed an intervention program combining medical hypnosis and music (Bissonnette et al., 2022; https://www.frontiersin.org/articles/10.3389/fpain.2022.926584/full).

Objectives and study design :

The main objective of this randomized control trial is to evaluate the efficacy of a personalized multimodal intervention program including hypnosis, music or their combination on composite score of pain, anxiety and unwellness as evaluated with the ESAS.

The secondary objectives are to assess :

* The evolution of distress and of each of the ESAS variables (pain, fatigue, nausea, depression, anxiety, sleepiness, appetite, unwellness, breathlessness) from pre-test to post-test compared with changes in these variables in the control group.
* The preference for the intervention modality (hypnosis, music or their combination).
* The feasibility of the experimentation in end-of-life palliative care at home.
* The experiential dimensions associated with music and hypnosis
* The subjective experience of the intervention.

Description of interventions :

The intervention program consists of a personalized multimodal intervention involving hypnosis and music. It offers each participant the option to receive (a) the hypnosis intervention presented as guided imagery, (b) the music intervention, or (c) a combination of (a) hypnosis (guided imagery) and (b) music. Each intervention is further personalized by integrating individually preferred imagery and/or music.

Recruitment and allocation procedure :

Adults (n = 40) in palliative home care receiving home support services from CIUSSS-NIM or CISSS-CA and meeting the inclusion criteria are eligible to participate in the project. The clinical team identifies participants who meet the selection criteria and asks them if they would like a visit from a member of the research team. During this visit, each participant is informed of the project and asked to sign the consent form. All participants then choose their preferred intervention modality (a. hypnosis, b. music or c. combination of hypnosis and music) before completing baseline measures including a socio-demographic questionnaire, the ESAS and a distress measure. Participants who choose an intervention with music (modalities a and c) are asked to identify pieces that they expect will generate positive emotions. Participants who choose guided imagery (modalities b and c) are asked to describe a pleasant place.

Participants are then stratified by gender and randomly assigned to the "experimental" group and the "control/waiting list" group. The distribution follows the order previously determined by a random table generated using an Excel function.

Two sessions are offered to the participants of the experimental group. During the sessions, a facilitator takes the pre-interventions measurements (see below), asks the participants to listen to the recorded intervention of 15 to 25 minutes by themselves while he/she waits outside the participant's home, and then comes back to fill in the post-intervention measurements (see below). Participants are also asked to report how they feel after each intervention and are given a brief semi-structured interview about their subjective experience.

Procedure in the two intervention sessions:

1. Measures (ESAS; Distress) (3-5 min)
2. Intervention Sessions (15-25 minutes)
3. Measures (ESAS; Distress; Experiential dimensions) (3-5 minutes)
4. Semi-structured interview about the subjective experience (2-5 min)

Participants in the control/waiting list group receive two control sessions following the same procedure as the experimental group but without receiving the intervention. During these control sessions, the same distress and ESAS measures are taken at 20-minute intervals. In the meantime, participants continue to perform their usual daily activities by themselves while the experimenter walk outside the participant's home.

Plan for each control session:

1. Measures (ESAS; Distress) (3-5 min)
2. Usual Daily Activities (20 min)
3. Measures (ESAS; Distress) (3-5 min)

After the two control sessions are completed, participants in the control/waiting list group receive two intervention sessions, following the same procedure as the experimental group. These supplementary sessions are not part of the main analysis design but will be examined as they provide additional pre-post intervention data.

Main objective:

To analyze the changes in the composite score of pain, anxiety, and unwellness between the beginning and the end of the sessions as a function of the group (control/waiting list vs. experimental), a mixed model repeated measures analysis procedures will be performed using SPSS software (GLM model). Data from all participants who completed at least one session will be retained and included in the analyses. Missing scores will be imputed by the model. We have also planned a sensitivity analysis taking into account the baseline level of the dependent variables, if there is a risk of a floor effect.

The data acquired in the additional sessions for the control group will be analysed separately and compared to the pre-post data obtained in sessions 1 and 2 in the same participants and in the experimental group.

The secondary objectives:

To assess the evolution of distress and of each of the ESAS variables of the experimental group from pre- to post-intervention and to evaluate the composite score for the intervention sessions in the control/ waiting list group we will apply a similar GLM model.

To assess the preference of the intervention modality (hypnosis, music, or hypnosis and music), we will count the frequency of selection of each intervention modality for all participants.

To assess the experiential aspects of the intervention, we will calculate the mean for each of the eight experiential dimensions.

To explore the subjective experience of the intervention, two open questions will be asked by the facilitator to inquire about the participant's current feeling and about their impression of change.

ELIGIBILITY:
Inclusion Criteria:

* End-of-life palliative care at home
* Between 30% and 79% on the Karnofsky Performance Index
* With adequate communication skills to complete the steps of the research
* With satisfactory or corrected hearing, as recommended by the caregiver.
* Severe neurocognitive or psychotic disorders

Exclusion Criteria:

* Severe neurocognitive or psychotic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in Composite pain, anxiety, and unwellness score | The posttest was administered 25 minutes after the pretest.
  Change in composite outcome score for pre-test to post-test for the experimental sessions compared with change in the control group. The composite score will be obtained by summing the pain (0-10), anxiety (0-10) and unwellness scores (0-10) from the Edmonton Symptom Assessment Scale. (ESAS)

SECONDARY OUTCOMES:
Changes in Pain levels | The posttest was administered 25 minutes after the pretest.
  Change in pain level, as assessed by the Edmonton Symptom Assesment Scale (ESAS) on a scale of 0 to 10.
Changes in Anxiety levels | The posttest was administered 25 minutes after the pretest.
  Change in anxiety level, as assessed by the Edmonton Symptom Assesment Scale (ESAS) on a scale of 0 to 10.
Changes in Unwellness levels | The posttest was administered 25 minutes after the pretest.
  Change in unwellness level, as assessed by the Edmonton Symptom Assesment Scale (ESAS) on a scale of 0 to 10.
Changes in Fatigue levels | The posttest was administered 25 minutes after the pretest.
  Change in fatigue level, as assessed by the Edmonton symptom assesment scale (ESAS) on a scale of 0 to 10.
Changes in Nausea levels | The posttest was administered 25 minutes after the pretest.
  Change in nausea level, as assessed by the Edmonton Symptom Assesment Scale (ESAS) on a scale of 0 to 10.
Changes in Depression levels | The posttest was administered 25 minutes after the pretest.
  Change in depression level, as assessed by the Edmonton Symptom Assesment Scale (ESAS) on a scale of 0 to 10.
Changes in Sleepiness levels | The posttest was administered 25 minutes after the pretest.
  Change in sleepiness level, as assessed by the Edmonton Symptom Assesment Scale (ESAS) on a scale of 0 to 10.
Changes in Appetite | The posttest was administered 25 minutes after the pretest.
  Change in appetite level, as assessed by the Edmonton Symptom Assesment Scale (ESAS) on a scale of 0 to 10.
Changes in Distress | The posttest was administered 25 minutes after the pretest.
  Change in distress level, as assessed by a Distress Thermometer on a scale of 0 to 10.
Preference of the intervention modality | At baseline
  The preference of the intervention modality by calculating the selection frequency (and the percentage) of each intervention across all participants.
Experiential dimensions | 1 week
  Ratings (0-10) obtained to characterize a) the participant's experience of mental absorption, b) change in perspective, c) experience of reminiscence, d) feeling of being understood, e) experience of transcendence, f) somatic experience, g) feeling of being in control
Feasibility of the study | Through study completion, an average of 1 year.
  To conduct the feasibility study, we will look at 1) the number of patients who have expressed initial interest in the study; 2) the number of participants recruited per month, 3) the proportion of patients who participate in the study out of the number of people in palliative home care for the entire experimental period, 4) the proportion of patients who complete the study.

OTHER OUTCOMES:
Subjective experience | 1 week
  Two open questions will be asked by the facilitator to inquire about the participant's current feeling (How do you feel?) and about their impression of change (What is different now compared to the beginning of the session?). The answers will be audio-recorded or noted by the facilitator.

CONTACTS AND LOCATIONS:
Overall Officials: Josiane Bissonnette, Ph.D, Principal Investigator — Laval University
Locations (2):
- Canada (2):
  - Ciusss-Nim, Montreal, Quebec
  - CISSS-CA, Saint-Georges, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bissonnette J, Dumont E, Pinard AM, Landry M, Rainville P, Ogez D. Hypnosis and music interventions for anxiety, pain, sleep and well-being in palliative care: systematic review and meta-analysis. BMJ Support Palliat Care. 2024 Jan 8;13(e3):e503-e514. doi: 10.1136/bmjspcare-2022-003551. PMID 35292511
- [Background] Bissonnette J, Pierre S, Duong ATJ, Pinard AM, Rainville P, Ogez D. Development of a Mixed Hypnosis and Music Intervention Program for the Management of Pain, Anxiety, and Wellbeing in End-of-Life Palliative Care. Front Pain Res (Lausanne). 2022 Jul 6;3:926584. doi: 10.3389/fpain.2022.926584. eCollection 2022. PMID 35875475